CLINICAL TRIAL: NCT00769405
Title: Phase III Study Evaluating the Use of Systemic Chemotherapy and Chemohyperthemia Intraperitoneal Preoperatively (CHIP) and After Maximum Resection of Peritoneal Carcinomatosis Originating With Colorectal Cancer
Brief Title: Systemic Chemotherapy With or Without Intraperitoneal Chemohyperthermia in Treating Patients Undergoing Surgery for Peritoneal Carcinomatosis From Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000595024; FRE-FNCLCC-ACCORD-15/0608; EUDRACT-2006-006175-20; EU-20847
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; peritoneal carcinomatosis
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Peritoneal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Diathermy

ARMS (2):
- Arm I (Experimental): Patients undergo surgery and receive standard systemic chemotherapy comprising leucovorin calcium IV followed by fluorouracil IV over 30 minutes. Systemic chemotherapy will continue for at least 6 months (before and after surgery). Patients also undergo CHIP comprising oxaliplatin intraperitoneally during surgery and hyperthermia for 30 minutes.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Procedure: hyperthermia treatment
- Arm II (Experimental): Patients undergo surgery and receive standard systemic chemotherapy comprising leucovorin calcium IV followed by fluorouracil IV over 30 minutes. Systemic chemotherapy will continue for at least 6 months (before and after surgery).
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium

INTERVENTIONS:
Drug: fluorouracil — Given IV
Drug: leucovorin calcium — Given IV
Drug: oxaliplatin — Given during surgery
  Arms: Arm I
Procedure: hyperthermia treatment — Given intraperitoneally during surgery
  Arms: Arm I

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as leucovorin, fluorouracil, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether systemic chemotherapy is more effective with or without intraperitoneal chemohyperthermia in treating patients with peritoneal carcinomatosis from colorectal cancer.

PURPOSE: This randomized phase III trial is studying systemic chemotherapy to see how well it works compared with or without intraperitoneal chemohyperthermia in treating patients undergoing surgery for peritoneal carcinomatosis from colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare overall survival of patients with peritoneal carcinoma of colorectal origin undergoing complete surgical resection and receiving systemic chemotherapy with versus without intraperitoneal chemohyperthermia.

Secondary

* Evaluate recurrence-free survival of these patients.
* Evaluate treatment toxicities.
* Determine morbidity from surgical complications.
* Determine prognostic factors of survival.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center, residual tumor status (R0/R1 vs R2 ≤ 1 mm), prior regimens of systemic chemotherapy (first vs ≥ second), and preoperative systemic chemotherapy for metastatic disease (yes vs no). Patients are randomized to 1 of 2 treatment arms.

All patients undergo maximal surgical resection of the tumor.

* Arm I: Patients receive standard systemic chemotherapy comprising leucovorin calcium IV followed by fluorouracil IV over 30 minutes. Systemic chemotherapy will continue for at least 6 months (before and/or after surgery). Patients must stop systemic chemotherapy at least 1 month before receiving intraperitoneal chemohyperthermia (CHIP). If bevacizumab is given as neoadjuvant therapy, then systemic chemotherapy must be discontinued 6 weeks before beginning CHIP. Patients undergo CHIP comprising oxaliplatin intraperitoneally during surgery and hyperthermia for 30 minutes.
* Arm II: Patients undergo surgery and receive standard systemic chemotherapy comprising leucovorin calcium IV followed by fluorouracil IV over 30 minutes. Systemic chemotherapy will continue for at least 6 months (before and after surgery).

Tumor markers (ACE and CA 19-9) are assessed at baseline, at 1 month after surgery, and then at follow-up visits.

After completion of study therapy, patients are followed at 1 and 3 months, every 3 months for 3 years, and then every 6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer

  * Peritoneal carcinoma extension ≤ 25 (Sugarbaker Index) (determined intraoperatively)

    * Planning to receive standard systemic chemotherapy

      * Chemotherapy for metastatic cancer should be initiated 3 months after surgery
    * No extraperitoneal metastases, including liver and lung metastasis
    * No carcinomatosis of other origin besides colorectal, in particular appendical carcinomatosis
* Macroscopically complete resection (R1) or surgical reduction of tumor to a residual thickness ≤ 1 mm (R2) is possible

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy > 12 weeks
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN
* Alkaline phosphatase ≤ 3 times ULN
* Creatinine ≤ 1.25 times ULN
* Eligible for surgery
* No peripheral neuropathy > grade 3
* Not pregnant or nursing
* No other cancer in the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix
* No inability to submit to follow-up medical testing for geographical, social, or psychological reasons
* Affiliated with a social security program
* Not deprived of liberty or under supervision

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemohyperthermia
* No concurrent participation in another study of first-line therapy for this cancer

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2008-02; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | until 3 years

SECONDARY OUTCOMES:
Recurrence-free survival | until 3 years
Toxicity by NCI CTCAE v.3.0 | until 5 years after surgery
Morbidity from surgical complications (abdominal, extra-abdominal, aplasia) | until 2 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Francois Quenet, MD, Principal Investigator — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (20):
- France (20):
  - Centre Paul Papin, Angers
  - Hôpital Antoine Béclère, Clamart
  - CHU Estaing, Clermont-Ferrand
  - Louis Mourier Hospital, Colombes
  - Hopital Du Bocage, Dijon
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Centre Leon Berard, Lyon
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Hopital de l'Archet CHU de Nice, Nice
  - Institut Curie, Paris
  - Hopital Lariboisiere, Paris
  - Hôpital Lariboisière, Paris
  - Hopital Tenon, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Jean Godinot, Reims
  - Hopital Universitaire Hautepierre, Strasbourg
  - Centre Hospitalier Regional de Purpan, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Quenet F, Elias D, Roca L, Goere D, Ghouti L, Pocard M, Facy O, Arvieux C, Lorimier G, Pezet D, Marchal F, Loi V, Meeus P, Juzyna B, de Forges H, Paineau J, Glehen O; UNICANCER-GI Group and BIG Renape Group. Cytoreductive surgery plus hyperthermic intraperitoneal chemotherapy versus cytoreductive surgery alone for colorectal peritoneal metastases (PRODIGE 7): a multicentre, randomised, open-label, phase 3 trial. Lancet Oncol. 2021 Feb;22(2):256-266. doi: 10.1016/S1470-2045(20)30599-4. Epub 2021 Jan 18. PMID 33476595